CLINICAL TRIAL: NCT04052412
Title: Biodistribution and Kinetics of 18F-AraG in Non-Small Cell Lung Cancer Patients Before and After Immunotherapy With and Without Radiation
Brief Title: Biodistribution and Kinetics of 18F-AraG in Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Collaborators: CellSight Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 4513
Record Dates: First submitted 2019-07-23; First posted 2019-08-09 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: This is a biodistribution and kinetics study looking at the uptake of 18F-AraG in non-small cell lung cancer patients in 3 different arms as follows:
  1. Non-small cell lung cancer undergoing immunotherapy without radiation therapy
  2. Non-small cell lung cancer undergoing immunotherapy with adjuvant radiation therapy
Who Masked: Care Provider
Masking Description: Physicians responsible for care are blinded to detailed study results to prevent any potential alterations to patient treatment. All treatment decisions are based on standard of care without regard for the biodistribution data collected from this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NSCLC with Immunotherapy without radiation (Experimental): The biodistribution and kinetics of the 18F-AraG compound will be assessed in non-small cell lung cancer patients undergoing immunotherapy without adjuvant radiation therapy
  Interventions: Drug: 18F-AraG
- NSCLC with Immunotherapy with radiation (Experimental): The biodistribution and kinetics of the 18F-AraG compound will be assessed in non-small cell lung cancer patients undergoing immunotherapy with adjuvant radiation therapy
  Interventions: Drug: 18F-AraG

INTERVENTIONS:
Drug: 18F-AraG — All arms of the study will receive an injection of 18F-AraG while on the PET imaging system. Following a 6 minute scan over the heart to acquire input function data, the patient will undergo a 1 hour multi-pass whole-body dynamic PET/CT acquisition to gather whole-body biodistribution data.

SUMMARY:
This study is to assess the biodistribution and kinetics of a novel T-cell imaging agent in non-small cell lung cancer patients undergoing immunotherapy with and without adjuvant radiation therapy. This study is assessing the change in kinetics that occurs in this patient population to better understand the distribution of this compound in patient disease circumstances.

DETAILED DESCRIPTION:
The overall goal of this project is to evaluate the ability of [18F]-AraG, a novel T-cell activation imaging biomarker, to measure T-cell activation before and after treatment with programmed death (PD) PD-1/PD-L1 inhibition and with PD-1/PD-L1 inhibition plus radiation therapy in NSCLC patients. Early preclinical and clinical studies have shown promise for immunotherapy treatments for several malignancies [1]. Immunotherapy is expected to grow in importance; however, it presents difficult challenges for response assessment. For instance, successfully treated tumors may actually increase in size after therapy due to inflammation and only later shrink [2]. RECIST criteria [3] designed to detect early effects of cytotoxic agents by size reduction, or the more recently proposed immune-related response criteria (irRC) [4] do not allow an early assessment of immunotherapeutic response since both depend on tumor size change. Furthermore, FDG PET is confounded by inflammatory effects causing hypermetabolism [5] [6]. Thus, it is imperative to develop new imaging and analysis protocols to evaluate immune-checkpoint blockade approaches. A method that evaluates T cell activation would permit an assessment of a basic first step in the process of assessing immunotherapy efficacy.

There are two main goals associated with this project. We propose to 1) assess the [18F]-AraG biodistribution and kinetics, in non-small cell lung cancer (NSCLC) tumor(s) and tumor draining lymph nodes on [18F]-AraG PET/CT imaging before and after 1 course of immunotherapy and 1 course of immunotherapy plus radiation 2) correlate (potential) change in [18F]-AraG uptake within the tumor(s) or tumor draining lymph nodes with clinical and pathologic response in patients treated with immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* This study is open to all adult subjects with histological confirmation of NSCLC enrolled in the parent protocol.
* Age 21 years of age or greater
* ECOG performance status of 0, 1, 2 or 3 at the time of enrollment.
* Patient with life expectancy ≥ 24 weeks from the time of screening to the study
* Ability to give informed consent

Exclusion Criteria:

* Patients with severe claustrophobia (patients with milder forms of claustrophobia that can be successfully allayed with oral anxiolytic therapy are allowed).
* Severe impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73 m2 and/or on dialysis.
* Pregnancy
* Breast Feeding an infant
* Unable to tolerate the expected radiation therapy prescription

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Biodistribution of 18F-AraG | Up to 90 minutes post injection of 18F-AraG
  Assessment of the distribution of 18F-AraG in patients with non-small cell lung cancer using activity concentration
Kinetics of 18F-AraG | Up to 90 minutes post injection of 18F-AraG
  Assessment of the rate of uptake using activity concentration of 18F-AraG in regions found to have significant AraG uptake

SECONDARY OUTCOMES:
Assessment of biodistribution and kinetics differences between study arms | 6 months
  Assessment of biodistribution and kinetics differences using activity concentration changes between patients undergoing immunotherapy with radiation and immunotherapy without radiation

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Osborne, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Medical Center, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Levi J, Lam T, Goth SR, Yaghoubi S, Bates J, Ren G, Jivan S, Huynh TL, Blecha JE, Khattri R, Schmidt KF, Jennings D, VanBrocklin H. Imaging of Activated T Cells as an Early Predictor of Immune Response to Anti-PD-1 Therapy. Cancer Res. 2019 Jul 1;79(13):3455-3465. doi: 10.1158/0008-5472.CAN-19-0267. Epub 2019 May 7. PMID 31064845
- [Background] Franc BL, Goth S, MacKenzie J, Li X, Blecha J, Lam T, Jivan S, Hawkins RA, VanBrocklin H. In Vivo PET Imaging of the Activated Immune Environment in a Small Animal Model of Inflammatory Arthritis. Mol Imaging. 2017 Jan 1;16:1536012117712638. doi: 10.1177/1536012117712638. PMID 28625080
- [Background] Ronald JA, Kim BS, Gowrishankar G, Namavari M, Alam IS, D'Souza A, Nishikii H, Chuang HY, Ilovich O, Lin CF, Reeves R, Shuhendler A, Hoehne A, Chan CT, Baker J, Yaghoubi SS, VanBrocklin HF, Hawkins R, Franc BL, Jivan S, Slater JB, Verdin EF, Gao KT, Benjamin J, Negrin R, Gambhir SS. A PET Imaging Strategy to Visualize Activated T Cells in Acute Graft-versus-Host Disease Elicited by Allogenic Hematopoietic Cell Transplant. Cancer Res. 2017 Jun 1;77(11):2893-2902. doi: 10.1158/0008-5472.CAN-16-2953. PMID 28572504
- [Background] Namavari M, Chang YF, Kusler B, Yaghoubi S, Mitchell BS, Gambhir SS. Synthesis of 2'-deoxy-2'-[18F]fluoro-9-beta-D-arabinofuranosylguanine: a novel agent for imaging T-cell activation with PET. Mol Imaging Biol. 2011 Oct;13(5):812-8. doi: 10.1007/s11307-010-0414-x. PMID 20838911